CLINICAL TRIAL: NCT01658384
Title: Cognitive Evolution in Tysabri Treated Multiple Sclerosis Patients
Acronym: CogMS
Status: Completed | Type: Observational
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: CogState Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNO-001
Record Dates: First submitted 2011-11-10; First posted 2012-08-07 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cognitive evolution, observational,MS: multiple sclerosis tysabri treated patients

SUMMARY:
This study is designed to evaluate the effect of Tysabri on cognition in multiple sclerosis (MS) patients. During a period of 24 months, the study will assess the evolution of cognitive function in Tysabri treated MS patients using the Symbol Digit Modalities Test (SDMT) and the CogState battery of tests.

DETAILED DESCRIPTION:
Tysabri reduces the relapse frequency, slows progression and preserves cognitive function as compared to placebo as per the AFFIRM trial. The benefit on relapse rate and progression appears to be sustained in longer-term studies such as STRATA. In clinical practice however despite a stable condition on the Expanded Disability Status Scale (EDSS) patients often complain of cognitive deterioration. It has yet to be shown that Tysabri will prevent cognitive deterioration after more than 2 years of treatment.

The Symbol Digit Modalities Test (SDMT) is a sensitive and validated test of cognition in MS. CogState offers a standardized battery of cognitive tests frequently used in clinical research in the fields of dementia and Parkinson's disease. The CogState battery of tests consisting of the Detection test (processing speed), Identification test (attention), One Back test (working memory), International Shopping List test (verbal learning) and the Groton Maze Learning test (reasoning and problem solving) will further confirm and validate the results of the Symbol Digit Modalities Test(SDMT) in MS patients as well as examine other cognitive parameters.

Together the above tests done prospectively can assess the evolution of cognitive function in Tysabri treated MS patients over the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis who are receiving Tysabri per indication and are willing and able to give an informed consent.

Exclusion Criteria:

* Patients who are depressed as per the Beck depression questionnaire at screening or at any time during the study.
* Patients with cognitive decline from causes other than MS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis who are receiving Tysabri per indication.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
SDMT CogState battery | 2 years
  Monthly cognitive assessments

CONTACTS AND LOCATIONS:
Overall Officials: François H Jacques, MD, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada